CLINICAL TRIAL: NCT05058482
Title: A Prospective, Multi-center, Randomized Parallel Controlled Study on the Safety and Effectiveness of the Non-adhesive Liquid Embolic System in the Embolization of Cerebral Arteriovenous Malformations
Brief Title: Non-adhesive Liquid Embolic System in the Embolization of Cerebral Arteriovenous Malformations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Hengruihongyuan Medical Technology Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nal01
Record Dates: First submitted 2021-09-24; First posted 2021-09-27 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2021-09

CONDITIONS: Intracranial Arteriovenous Malformations
Keywords: Non-adhesive Liquid Embolic System
MeSH Terms: conditions — Intracranial Arteriovenous Malformations | interventions — Embolic Protection Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-adhesive Liquid Embolic System(NALES) (Experimental)
  Interventions: Device: embolism
- Onyx Liquid Embolic System& Marathon Flow Directed Micro Catheter (Active Comparator)
  Interventions: Device: embolism

INTERVENTIONS:
Device: embolism — Cerebral arteriovenous malformation embolism

SUMMARY:
This clinical trial is to verify the safety and effectiveness of the Non-adhesive Liquid Embolic System(NALES) produced by Suzhou Hengrui Hongyuan Medical Technology Co., Ltd. in the process of clinical use to support the application of the National Medical Products Administration ( NMPA) product registration approval.

DETAILED DESCRIPTION:
A prospective, multicenter, randomized controlled trial was used in this study. Onyx Liquid Embolic System and Marathon Flow Directed Micro Catheter, which were registered and marketed in China and had good effect in the industry, were selected as the control devices. Subjects requiring cerebral arteriovenous malformation embolization were selected to participate in the trial based on pathological conditions and inclusion/exclusion criteria, and the use of test products or control products was determined based on central randomized results. Imaging data involving the main evaluation criteria were evaluated uniformly by the blind evaluators of the leading unit, so as to reduce the bias caused by subjective factors of different evaluators.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, no gender limit.
2. The patient was diagnosed as cerebral arteriovenous malformation .
3. The patient had no history of bAVM treatment, including intervention, surgery or radiotherapy .
4. Spetzler Martin, grade I-IV .
5. The patient voluntarily signed the informed consent.

Exclusion Criteria:

1. History of heparin allergy.
2. The patient is allergic to contrast media.
3. Severe hepatic and renal insufficiency (serum creatinine ≥1.5 times the upper limit of normal value, alanine aminotransferase ≥3 times the upper limit of normal value, aspartate aminotransferase ≥3 times the upper limit of normal value).
4. Patient has irreversible coagulopathy (INR > 1.5).
5. Intracranial hemorrhage 1 week before treatment.
6. MRS ≥4 due to neurological dysfunction.
7. Patients with planned malformation resection after embolization.
8. Blood flow related aneurysms of supplying artery that need to be treated by other methods.
9. Complicated with severe cerebral artery stenosis.
10. Brain tumors that require recent surgery.
11. Complicated with proliferative cerebrovascular disease.
12. Pregnant or lactating women.
13. Participants who have participated in other clinical trials within the last 3 months and failed to reach the end point.
14. The number of embolism is expected to be greater than or equal to 4 times during the study period (within 1 year).
15. Subjects deemed unsuitable for this study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-12-02 (Actual); Primary Completion 2023-10-17 (Estimated); Study Completion 2024-10-17 (Estimated)

PRIMARY OUTCOMES:
Effective embolization rate of malformed masses | Immediately after surgery
  Number of effective embolization subjects / Total number of subjects x 100%.Definition of effective embolization : Postoperative DSA angiographic malformation volume decreased ≥50%. Volume of malformed groups = length × width × height /2.

SECONDARY OUTCOMES:
MRS score | 1,6,12months after surgery
  MRS refers to the modified Rankin scale, which is used to measure the neurological recovery of patients after stroke. It has a scale of zero to six. The higher the score, the worse the neurological function. MRS scores were collected at 1, 6 and 12 months after the operation before discharge .
Technical success rate | Immediately after surgery
  Success is represented by the ability to reach the lesion and embolize the malformed mass of the intended target, followed by successful catheter withdrawal from the body
Catheter performance evaluation | Immediately after surgery
  1. The ability of the catheter to reach the lesion .
  2. The catheter has broken at the tip and perforated.
  3. Intravascular complications associated with catheters occurred.
  4. Degree of difficulty in tube withdrawal
  5. Catheter jam

OTHER OUTCOMES:
Incidence of major adverse events related to device or surgical procedures within 1 month after surgery | 1 month after surgery
  Major adverse events related to instrumentation or surgical procedures within 1 month after surgery: bleeding during embolization, catheter indwelling, bleeding after embolization, symptomatic cerebral infarction, and edema.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nan Fang Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjng Drum Tower Hospital, Nanjing, Jiangsu
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Huashan Hospital ,Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang